CLINICAL TRIAL: NCT04245423
Title: The Whole Health Study: Collaborative Care for OUD and Mental Health Conditions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, David Mandell, Kenneth E. Appel Professor and Director, Penn Center for Mental Health, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UF1MH121944 (NIH)
Record Dates: First submitted 2020-01-25; First posted 2020-01-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Opioid-use Disorder; Mental Health Conditions
Keywords: Opioid-use disorder; Depression; Anxiety; Post-traumatic stress disorder; Collaborative Care
MeSH Terms: conditions — Opioid-Related Disorders; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Augmented Usual Care (AUC) (Active Comparator): If not already waivered, PCPs will be trained and waivered to treat OUD with medications. Almost all practices have hired mental health clinicians, equivalent to the care managers in the investigators' collaborative care model, to treat mild and moderate depression and anxiety. These clinicians typically are licensed clinical social workers; a few are nurses or psychologists. No care managers have received systematic training in treating patients with OUD. The clinicians will retain their role and continue to treat and monitor patients with mental health conditions in these practices. Other than that, the research team will provide no support to the PCP or practice staff. However, an addiction psychiatrist is available for consultation for OUD. Patients are informed that the primary care practice provides both OUD and mental health treatment and are referred back to their provider for referral or to schedule care. A list of available community resources are available to the patient.
  Interventions: Behavioral: Augmented Usual Care
- Collaborative Care (CC) (Experimental): CC condition includes the following elements:
  1. Personnel trained to assist with scheduling, reminders and referrals;
  2. PCP trained and waivered to provide evidence-based pharmacotherapy for OUD;
  3. Addictions psychiatrist with collaborative care expertise to provide treatment consultation and supervision in both OUD and mental health issues;
  4. A care manager trained in evidence-based interventions for individuals with OUD and psychiatric disorders, who provides care in the primary care practice as part of the collaborative care team;
  5. Measurement-guided care and treat-to-target practices, using validated measures of substance use, depression, anxiety as well as measures of adherence and side effects;
  6. Electronic and in-person systematic communication regarding patient care among team members, facilitated by the electronic health record; and
  7. Shared patient-provider decision making.
  Interventions: Behavioral: Collaborative Care for Opioid Use Disorders and Mental Health Conditions
- Collaborative Care + Certified Recovery Specialist (CC+) (Experimental): In addition to the collaborative care model described above, patients in the CC+ condition will have access to a Certified Recovery Specialist (CRS) to assist with treatment engagement and retention. A CRS is a person in the community who is in recovery and may share similar experiences and barriers that participants have faced. They will work with participants as a peer to help them coordinate information and needs with their providers. The CRS will take participants to their PCP appointments and any other appointments that they may have to help them engage and stay in care to remain healthy. They will also provide education and help participants work on their recovery goals. They will identify and support linkages to community resources and help participants identify barriers to full participation in their recovery and develop strategies to overcome those barriers.
  Interventions: Behavioral: Collaborative Care for Opioid Use Disorders and Mental Health Conditions Plus Certified Recovery Specialists

INTERVENTIONS:
Behavioral: Collaborative Care for Opioid Use Disorders and Mental Health Conditions — CC is delivered using the investigators' Foundations for Integrated Care model. The first line pharmacotherapy is buprenorphine-naloxone. The second line pharmacotherapy included is extended-release injectable naltrexone. Pharmacotherapy is accompanied by brief problem-solving therapy, cognitive-behavioral therapy, and/or motivational interviewing. The primary care physician, in consultation with the addictions psychiatrist and care manager, also will provide psychotropic medications for psychiatric disorders. In-person and telephone visits consist of the care manager carrying out intervention activities over 6 months. Visits are at baseline (90-minute intake appointment), home or office induction when in moderate opiate withdrawal if buprenorphine is prescribed, twice a week for two weeks with telephone calls in between visits, then weekly, and when stable once a month. There will be a final visit at 6 months. The intervention includes routine collection of urine drug screens.
  Arms: Collaborative Care (CC)
Behavioral: Augmented Usual Care — If not already waivered, PCPs will be trained and waivered to treat OUD with medications. All practices will have mental health clinicians to treat mild psychiatric disorders. Other than that, the research team will provide no support to the PCP or practice staff. However, an addiction psychiatrist is available for consultation for OUD.
  Arms: Augmented Usual Care (AUC)
Behavioral: Collaborative Care for Opioid Use Disorders and Mental Health Conditions Plus Certified Recovery Specialists — This intervention includes the Collaborative Care Intervention plus Certified Recovery Specialist to assist with treatment engagement and retention.
  Arms: Collaborative Care + Certified Recovery Specialist (CC+)

SUMMARY:
Collaborative care for mental health is increasingly common, but most primary care practices have not embraced similar models for opioid use disorder (OUD). This study will refine and test a collaborative care model for patients with opioid use disorder (OUD) and depression, anxiety or post-traumatic stress disorder (PTSD) in primary care. We also will examine clinician and practice characteristics associated with successful implementation and the cost effectiveness of different care models.

DETAILED DESCRIPTION:
This research aims to refine and rigorously test a collaborative care model for patients with opioid use disorder (OUD) and depression, anxiety disorder, or post-traumatic stress disorder (PTSD) in primary care. The investigators will also examine clinician and practice characteristics associated with successful implementation and the cost effectiveness of different care models. The primary aims of this proposal are: (1) Rapidly prototype and test our collaborative care models to optimize them for implementation at the University of Pennsylvania Health System (UPHS) primary care clinics for the treatment of individuals with co-occurring mental health problems and opioid use disorder (OUD); (2) Conduct a randomized clinical trial (RCT) among 1,185 primary care patients aged 18 years and older with OUD and depression, anxiety or PTSD. Patients will be randomized to one of three conditions:

a) Augmented Usual Care (AUC), which consists of a primary care physician (PCP) waivered to prescribe buprenorphine, a mental health care manager, and an addiction psychiatrist to consult on Medication-Assisted Treatment (MAT); b) Collaborative Care (CC), which consists of a waivered PCP, a mental health care manager who receives OUD training, and a psychiatrist who provides telephonic consultation for OUD and mental health; or c) Collaborative Care Plus (CC+), which consists of all the elements of CC, plus a Certified Recovery Specialist (CRS) to help with patient engagement in treatment and retention in care;

(3) Measure clinician- level factors associated with implementation of each component and metrics of fidelity and reach, our primary implementation outcomes of interest; and (4) Assess the costs to primary care practices of implementing and delivering AUC, CC and CC+ and the change in total healthcare costs associated with the implementation. Successful completion of the proposed study will provide definitive evidence regarding the most parsimonious set of elements of integrated collaborative care required to maximize outcomes for individuals with OUD and psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older;
2. a diagnosis of opioid use disorder using DSM-5 criteria within the last 12 months OR have taken medication for opioid use disorder (MOUD) within the last 12 months;
3. agree to receive medication for opioid use disorder at the primary care site (the first line pharmacotherapy is buprenorphine-naloxone and the second line pharmacotherapy will include extended-release injectable naltrexone);
4. meet criteria for depression, anxiety (panic disorder, social anxiety disorder, obsessive-compulsive disorder, or generalized anxiety disorder), or PTSD;
5. able to communicate in English; and
6. willing to give informed consent.

Exclusion Criteria:

1. acutely suicidal and needs immediate hospitalization, manic or psychotic (patients will not be randomized and PI or study physician covering for PI will be notified immediately); and
2. lack of a phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 567 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in opioid use based on self-reported | Baseline and monthly for 6 months
  Modified Timeline Followback
Change in opioid use based on toxicology | Baseline and monthly for 6 months
  Urine Drug Screens
Change in psychiatric symptoms - Depression | Baseline and monthly for 6 months
  Patient Health Questionnaire (PHQ-9); range is 0-27 with higher scores demonstrating worse outcomes
Change in psychiatric symptoms - Anxiety | Baseline and monthly for 6 months
  Generalized Anxiety Disorder Screener (GAD-7); range is 0-21 with higher scores demonstrating worse outcomes
Change in psychiatric symptoms - Post-traumatic Stress Disorder | Baseline and monthly for 6 months
  Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5); range is 0-80 with higher scores demonstrating worse outcomes

SECONDARY OUTCOMES:
Change in Illicit use of other drugs besides opioids (e.g. benzodiazepines, cocaine) | Baseline and monthly for 6 months
  Modified Timeline Followback
Change in medication adherence | Baseline and monthly for 6 months
  Self-report
Treatment retention | 6 months
  Measured as the time to dropout (from both OUD and mental health treatment using clinic records)
Rate of Mortality | 6 months
  Assessed through death records

CONTACTS AND LOCATIONS:
Overall Officials: David Mandell, ScD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Center for Primary Care, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Harris RA, Campbell K, Calderbank T, Dooley P, Aspero H, Maginnis J, O'Donnell N, Coviello D, French R, Bao Y, Mandell DS, Bogner HR, Lowenstein M. Integrating peer support services into primary care-based OUD treatment: Lessons from the Penn integrated model. Healthc (Amst). 2022 Sep;10(3):100641. doi: 10.1016/j.hjdsi.2022.100641. Epub 2022 Jul 2. PMID 35785613
- [Derived] Harris RA, Mandell DS, Kampman KM, Bao Y, Campbell K, Cidav Z, Coviello DM, French R, Livesey C, Lowenstein M, Lynch KG, McKay JR, Oslin DW, Wolk CB, Bogner HR. Collaborative care in the treatment of opioid use disorder and mental health conditions in primary care: A clinical study protocol. Contemp Clin Trials. 2021 Apr;103:106325. doi: 10.1016/j.cct.2021.106325. Epub 2021 Feb 22. PMID 33631356

DOCUMENTS (1):
  • Informed Consent Form (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/23/NCT04245423/ICF_000.pdf